CLINICAL TRIAL: NCT01527240
Title: Cyclosporin A Combined to Intravenous Thrombolysis. Multicenter Randomized Placebo-controlled
Brief Title: Neuroprotection Impact of Cyclosporin A in Cerebral Infarction
Acronym: CsAStroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008.544
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2012-01

CONDITIONS: Stroke
Keywords: Volume of cerebral infarction; Stroke; CsA; NIHSS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciclosporin A (Experimental): Injection of 50 mg / ml IV infusion. 5 ml ampoules (250 mg of ciclosporin)
  Interventions: Drug: Ciclosprin A
- Placebo (Placebo Comparator): Injectable Saline Solution.
  Interventions: Drug: Injectable Saline Solution.

INTERVENTIONS:
Drug: Ciclosprin A — The dose in this study was 2 mg / kg, administered within 15 min after beginning of thrombolysis. The treatment of the study consists of a single bolus injection. This dose was chosen according to the results of tolerance in myocardial infarction and unknown pharmacodynamic and safety data
  Arms: Ciclosporin A
Drug: Injectable Saline Solution. — Saline Solution is administered once 15 min after thrombolysis.
  Arms: Placebo

SUMMARY:
The main objective of this study is to determine whether a single injection of CsA after intravenous thrombolysis can significantly decreased the volume of cerebral infarction at day 30 ± 15 assessed with Flair MRI.

Secondary objectives are to determine whether a single injection of CsA after intravenous thrombolysis is safe and effective regarding to death and disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years and <85 years
* Male or female,
* Patients with cerebral infarction of less than 4:30H,
* NIHSS score between 6 and 18
* Identification of a carotid artery occlusion in the territory in MRI
* Consent of participation signed by the patient or, if it is unable to give the family or someone you trust if it is present.
* Patient beneficiary of a social security system.

Exclusion Criteria:

* Known hypersensitivity to cyclosporin A or castor oil, polyoxyethylene
* Patient in St. John's wort, stiripentol, bosentan or rosuvastatin
* History of immunosuppression recent (<6 months): cancer, lymphoma, positive serology for HIV, hepatitis, ...
* Known hepatic (prothrombin time <50%)
* Patients treated with sulfonylureas or nicorandil
* Patients treated with dopamine, adrenaline, noradrenaline or isoprenalin
* Uncontrolled hypertension defined as systolic blood pressure greater than 185mm Hg and a diastolic pressure above 110 mmHg,
* Cardiogenic shock defined by systolic blood pressure below 80 mm Hg
* Contraindication to thrombolysis: History of AIC in the three months history of intracranial hemorrhage, neoplasm, subarachnoid hemorrhage, arteriovenous malformation
* Presumption of septic embolism or aortic dissection or pericardial effusion.
* Recent biopsy or surgery within 3 months
* Head injury less than 3 months
* Known bleeding diathesis, taking anticoagulants with INR> 1.2
* Hypoglycemia (blood glucose below 0.5 mmol / l)
* Known renal, creatinine greater than 130 Mu / L
* Recent Lumbar puncture <7days
* Conditions prior psychiatric or neurological deficit does not allow objective analysis of disability
* History of ischemic stroke or hemorrhagic
* History of epilepsy and taking antiepileptic
* Exclusion criteria Imaging
* Structured hypodensity scanner compatible with recent ischemic stroke
* Hematoma
* Other lesions (tumor or inflammatory cerebral venous thrombosis)
* The scanner Contraindications: allergy to iodine or major renal creatinine> 130μl or MRI referred to above
* Women of childbearing age, pregnant or not recognized effective contraception
* Patients in the measure of legal protection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
to determine whether a single injection of CsA after intravenous thrombolysis significantly decreased the volume of cerebral infarction at day 30 ± 15 in the T2-weighted Flair MRI. | at day 30 ± 15 in the T2-weighted Flair MRI.
  Volume of cerebral infarction at day 30 ± 15 in the T2-weighted MRI Flair will be measured by manuel contouring by two independent radiologists uninformed of clinical and therapeutic data and therapeutic

SECONDARY OUTCOMES:
to determine whether a single injection of CsA after intravenous thrombolysis, is well tolerated and reduces deaths and disability in patients. | on day 1, J7, J30, J90
  Secondary endpoints include clinical scores: NIHSS , mRS, Death, SAE (within neurological worsening of more than 4 points on the NIHSS).

CONTACTS AND LOCATIONS:
Overall Officials: Norbert NIGHOGHOSSIAN, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Nighoghossian N, Berthezene Y, Mechtouff L, Derex L, Cho TH, Ritzenthaler T, Rheims S, Chauveau F, Bejot Y, Jacquin A, Giroud M, Ricolfi F, Philippeau F, Lamy C, Turc G, Bodiguel E, Domigo V, Guiraud V, Mas JL, Oppenheim C, Amarenco P, Cakmak S, Sevin-Allouet M, Guillon B, Desal H, Hosseini H, Sibon I, Mahagne MH, Ong E, Mewton N, Ovize M. Cyclosporine in acute ischemic stroke. Neurology. 2015 Jun 2;84(22):2216-23. doi: 10.1212/WNL.0000000000001639. Epub 2015 May 6. PMID 25948727